CLINICAL TRIAL: NCT05484609
Title: Examining Access to Primary Care for People With Opioid Use Disorder: a Randomized Controlled Audit Study
Brief Title: Access to Primary Care for People With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Sheryl Spithoff, Scientist and Clinician Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 410012447
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Access to Primary Care
Keywords: primary care; access to health care; opioid use disorder; addictions; health services
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: 1:1 allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OUD scenario (Experimental)
  Interventions: Other: OUD scenario
- Diabetes scenario (Active Comparator)
  Interventions: Other: Diabetes scenario

INTERVENTIONS:
Other: OUD scenario — The patient actor will make unannounced phone calls to family physicians asking for a new patient appointment. The patient actor will play the role of a patient with opioid use disorder undergoing methadone treatment with an addiction physician.
  Arms: OUD scenario
Other: Diabetes scenario — The patient actor will make unannounced phone calls to family physicians asking for a new patient appointment. The patient actor will play the role of patient with diabetes in treatment with an endocrinologist.
  Arms: Diabetes scenario

SUMMARY:
Background: Access to high quality primary care is essential for health, particularly for vulnerable populations. Research indicates, however, that people with opioid use disorder (OUD), are less likely than others to have a primary care provider. The reasons are unclear, but may be related to patient factors, system barriers and provider factors, including discrimination.

Research goal: Our primary goal is to determine if discrimination by primary care physicians plays a role in poor access to primary care for those in treatment for OUD. The answers will help researchers and policy-makers find ways to improve access to primary care for this vulnerable population.

Research question: Are people in treatment for OUD less likely to be offered a new patient appointment with a physician compared to those in treatment for diabetes? Overall study design: In this randomized controlled trial (RCT), the investigators will make unannounced phone calls to primary care physicians' practices to ask for a new patient appointment. Physicians will be randomly assigned to one of two clinical scenarios: a patient with diabetes, or a patient in treatment for OUD. Our outcome measure is an unconditional offer of a new patient appointment with the physician contacted or with another physician at the same practice. In an secondary analysis the investigators will determine the impact of physician gender, years in practice, rurality and model of care on offers of a new patient appointment.

Participants: Randomly-selected primary care physicians in Ontario. Data analysis methods: The investigators will use chi-squared test and logistic regression to determine if there is a statistically and clinically significant difference in the proportions of offering a new patient appointment between the two clinical scenarios.

DETAILED DESCRIPTION:
Study context

According to the World Health Organization (WHO) primary health care is a "highly effective and efficient way to address the main causes and risks of poor health and wellbeing today" (1). Primary care is particularly important for vulnerable populations as it appears to mitigate effects from factors like low socioeconomic status (2-4). This appears to be true for those with opioid use disorder (OUD): in previous work, enrolment to a primary care physician was associated with higher rates of cancer screening and diabetes monitoring for those in treatment for OUD (5).

In universal health care systems, like Canada's, everyone is entitled to primary health care, regardless of health conditions or financial status. Our previous work, however, indicates that Ontarians in treatment for OUD are less likely to have access to primary care than others. Only 43% of people in treatment for OUD were enrolled with a primary care physician compared to 73% of matched controls (5). Our findings are consistent with an American study that reported poor access to primary care for those in treatment for OUD (6). These findings are concerning. Not only are those with OUD a vulnerable population with complex health needs, their numbers are also growing. OUD currently affects 15.5 million people worldwide (7), with Canada and the United States (U.S.) having the highest burden of disease (8).

Barriers to primary care for those with OUD have been poorly studied. Patient factors, such as difficulty attending appointments, and system barriers, like transportation costs, may affect access (9). Provider factors appear to play a role as well. A qualitative interview study in Ontario found that provider discrimination and stigma towards those with substance use disorder presented a barrier to accessing primary care (9). Other studies support this finding, showing that many providers, just like the general public, have stigma towards those with substance use disorder (10,11). It is possible that negative attitudes lead providers to discriminate against people with OUD when deciding whether to offer a new patient appointment.

Study rationale and goal

Our study goal is to determine if discrimination by physicians is a barrier to accessing primary care for those with OUD.

Research questions

1. Are people in treatment for OUD less likely to be offered a new patient appointment compared to people in treatment for diabetes?
2. What is the impact of physician gender, years in practice, rurality and model of care on offers of a new patient appointment?

Methods

The investigators will conduct a randomized controlled trial (RCT), using a similar approach to Olah et al that looked at access to primary care for those of low socio-economic status (14). They will make unannounced phone calls to primary care physicians in Ontario asking for a new patient appointment. Physicians will be randomly assigned to one of two clinical scenarios: a patient with diabetes treated by an endocrinologist, or a patient with OUD prescribed methadone by an addiction physician. In the secondary exploratory analyses, the investigators will also assess the impact of the model of care (team vs not), gender, rural vs urban, and years in practice.

Population The investigators will use information on the College of Physicians and Surgeon of Ontario (CPSO) website to identify all physicians in Ontario who have an active, independent, unrestricted practice with a self-reported speciality in family medicine (20).

Sample size calculation The objective of our study is to compare the proportion of patients offered a new patient appointment in each of the arms of the study. Our team consensus was that a 10% difference in the proportion of new patient appointments would be clinically meaningful. In a similar study design, Olah et al found that 23.5 % of those with diabetes were offered an appointment from a physician in Ontario (14). For our sample size calculation, the investigators assumed that 23% of those with diabetes and 13% of those in treatment for OUD would be offered a new appointment. At 80% power, 5% type-1 error level, to detect 10% difference in the proportion of new appointments offered between opioid (13%) and diabetes (23%) groups, would require 231 physicians with each scenario. However, previous studies using this approach found that up to one third of physicians were excluded at the time of making the phone call (because physician worked in a walk-in clinic or had a practice that was not primary care; or because of no response after five phone calls) (14,18). Therefore, the study should include 308 physicians in each arm.

To create our sample, the investigators will create a database using publicly-available information on the CPSO website. They will include all physicians who have an active, unrestricted, independent practice with speciality in Family Medicine. They will also record the physician's address(es), postal code, phone number(s), date of registration for independent practice and gender in our database. Physicians will only be identified in the database by a unique identifier. All these data items are collected by the CPSO. They will then group the physicians by primary practice address and then randomly select (using a random number generator), one physician from the list of physicians who work at the same site. The investigators will exclude other physicians from the same practice address.They will then use a random number generator to randomly select a statistical determined sample of physicians. We will randomly assign them to one of two clinical scenarios: a patient with diabetes treated by an endocrinologist, or a patient with OUD prescribed methadone by an addiction physician.

Scenarios The investigators will train a research assistant (RA) in the clinical scenario and pilot-test the interaction with a simulated receptionist giving different responses (see Appendix 1: Sample Script). To reduce confounding, they will have the same RA make all the phone calls. The RA will contact each physician to request an appointment, for one of the two clinical scenarios. The investigators will exclude physicians at the time of making the phone call if the physician's receptionist reports that the clinic is a walk-in, or that the physician does not offer primary care (14). They will also exclude practices at the time of making the call if they request an in person visit or health card number prior to making an offer of a new patient appointment. The investigators will attempt to reach a physician up to five times over a six-week period. For offices with voicemail, they will leave a message with the script but continue to make up to five phone calls to speak with someone in person. The investigators will accept call-backs up to six weeks after the initial phone call. They will exclude practices where they are not able to speak to anyone or leave a voicemail after five phone calls. They will only request an appointment once from a physician. If the physician's clinic offers an appointment, they will call the next day and cancel it. The investigators will continue sampling until they reach our target number of physicians.

Data analysis The investigators will use descriptive statistics to report on the population. To answer our research question, they will compare the proportion of patients offered a primary care appointment (a binary outcome) across the randomized groups. They will use chi-squared test and logistic regression to determine if there is a statistically and clinically significant difference in the proportions of offering a new patient appointment between the two clinical scenarios.

The investigators expect groups to be balanced on measured and unmeasured confounding variables. Nonetheless, they will investigate the distribution of measured variables across the two groups. If they observe imbalances, they will estimate the adjusted impact on the likelihood of being offered a new appointment, after controlling for possible confounding factors.

For our secondary analyses the investigators will use Fisher Exact test and two sample Wilcoxon test to assess if pre-specified subgroups: physician gender (male vs. female); practice location (rural < 50,000 vs. urban practice setting > 50,000); years in clinical practice, and practice model (team-based vs. not) affected the likelihood that a patient would receive an unconditional offer of a new patient appointment.

The investigators expect groups to be balanced on measured and unmeasured confounding variables. Nonetheless, they will investigate the distribution of measured variables across the two groups. If they observe imbalances, they will estimate the adjusted impact on the likelihood of being offered a new appointment, after controlling for possible confounding factors.

For our secondary analyses the investigators will use Fisher Exact test and two sample Wilcoxon test to assess if pre-specified subgroups: physician gender (male vs. female); practice location (rural < 50,000 vs. urban practice setting > 50,000); years in clinical practice, and practice model (team-based vs. not) affected the likelihood that a patient would receive an unconditional offer of a new patient appointment.

ELIGIBILITY:
Inclusion Criteria:

* physicians with an active, unrestricted, independent practice in Ontario with a self-reported specialty in Family Medicine

Exclusion Criteria:

* physicians with restricted practices (e.g., could not prescribe opioids)
* physician not in independent practice (i.e., physicians in training)
* physicians whose practice address is in a community with a population less than 10,000, unless they are close (less than 50km) to a community with a population greater than 20,000.
* physicians who do not provide primary care
* physicians who require a health card number prior to offering a new patient appointment
* physicians who require an in person visit prior to offering a new patient appointment
* physicians who we are unable to reach after five phone calls and do not have voicemail
* physicians who work at same practice address as another randomly-selected physician included in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an offer of a new patient appointment | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl M Spithoff, MD MSc, Principal Investigator — Women's College Hospital
Locations (1):
- Province of Ontario, Ontario, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Spithoff S, Mogic L, Hum S, Moineddin R, Meaney C, Kiran T. Examining Access to Primary Care for People With Opioid Use Disorder in Ontario, Canada: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2233659. doi: 10.1001/jamanetworkopen.2022.33659. PMID 36178686